CLINICAL TRIAL: NCT01533389
Title: A 4-week, Double-blind, Randomized, Comparative and Multi-center Clinical Trial to Evaluate the Efficacy and Safety of Silodosin in the Treatment of Natural Expulsion in Patients With Ureteral Stones.
Brief Title: Efficacy and Safety of Silodosin in the Treatment of Natural Expulsion in Patients With Ureteral Stones
Acronym: STONE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: JW Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CWP-SDS-404
Record Dates: First submitted 2012-02-06; First posted 2012-02-15 (Estimated); Last update posted 2013-11-20 (Estimated); Status verified 2013-11

CONDITIONS: Ureteral Stone
MeSH Terms: conditions — Ureterolithiasis | interventions — silodosin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Silodosin (Experimental): 8mg QD
  Interventions: Drug: Silodosin
- Placebo (Placebo Comparator): 8mg QD
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Silodosin — Drug: silodosin dosage form : capsule dosage : placebo 4mg*2 (8mg) frequency and duration : QD, 4weeks
  Arms: Placebo
  Arms: Silodosin
Drug: Placebo — dosage form : capsule dosage : placebo 4mg*2 (8mg) frequency and duration : QD, 4weeks
  Arms: Placebo

SUMMARY:
A lower ureteral calculus, which measures 5 millimeters and less, may be easily expelled by symptomatic therapy. Actually, it has about a 50% chance of successful expulsion.

However, a complication such as urinary tract infection or hydronephrosis or persistent pain may occur before it is expelled. Thus, it is imperative to minimize the occurrence of complications in the process of expectant treatment and also to reduce the time required to expel calculi.

Pharmacotherapy is to relieve ureteral obstruction and thus to expel urinary calculi easily.

This clinical trial is to evaluate the efficacy of silodosin, a selective α1A-blocker, on calculous expulsion in expectant treatment for patients with lower and mid ureteral calculi.

DETAILED DESCRIPTION:
Lower and mid ureteral calculi, accounting for approximately 70% of ureteral calculi, has a high chance of successful treatment thanks to ureteroscopic lithotripsy or extracorporeal shock wave lithotripsy (ESWL)1-3), but at the same time have problems of postprocedural complications and high expenses4). A lower ureteral calculus, which measures 5 millimeters and less, may be easily expelled by symptomatic therapy. Actually, it has about a 50% chance of successful expulsion5). However, a complication such as urinary tract infection or hydronephrosis or persistent pain may occur before it is expelled. Thus, it is imperative to minimize the occurrence of complications in the process of expectant treatment and also to reduce the time required to expel calculi.

It has been recently reported that pharmacotherapy is adhibited to the expulsion of urinary calculi and the relief of pain. The migration of ureteral calculi is influenced by both the calculus and the ureter. In the case of the calculus, size, shape, number and location influence it. In regard to the ureter, it is significantly influenced by the cramp of the ureteral smooth muscle, the edema of the ureteral submucosa, the pain caused by the calculus and the activities of adrenoreceptors6).

Pharmacotherapy is to relieve ureteral obstruction and thus to expel urinary calculi easily. Ureteral obstruction, caused by urinary calculi, obtunds ureteral peristalsis but strengthens ureteral contraction, which may cause urinary retention or regurgitation7-8). In this connection, studies have been conducted as to methods to reduce abnormal urinary reaction caused by urinary calculi and to smoothen uroflow. Currently, hormone drugs including hydroxyprogesterone, prostaglandin synthetase inhibitors, calcium-channel antagonists, α1-blockers and steroid drugs are used to expel urinary calculi and to suppress pain. The guidelines on urinary calculi, drawn up in 2007, recommend using α-blockers as they are superior to other drugs in efficacy9-12).

The drug to be used in this clinical trial, silodosin, was registered under the proprietary name of 'THRUPAS® Capsule 4mg' and is being marketed after being authorized by Korea Food and Drug Administration (FDA), which selectively acts on the α1A-adrenoreceptor.

This clinical trial is to evaluate the efficacy of silodosin, a selective α1A-blocker, on calculous expulsion in expectant treatment for patients with lower and mid ureteral calculi.

ELIGIBILITY:
Inclusion Criteria:

* Males or female patients aged 20 and over
* Patients having ureteral calculi located mid or lower ureter on abdominal radiograms or excretory urograms or non-enhanced computed tomograms.
* Patients whose calculi measure 10 millimeters and less.
* Patients who voluntarily decided to take part in this clinical trial and gave written consent.

Exclusion Criteria:

* Patients who do not want to undergo expectant treatment
* Female patients who are pregnant or nursing
* Patients with febrile urinary tract infection or severe hydronephrosis or ulcerative diseases or hypotension.
* Patients with severe hepatic dysfunction(e.g. hepatic failure, hepatic cirrhosis, icterus, hepatoma)
* Patients who take α-blocker or α/β-blockers or calcium-channel blockers or steroid drugs
* Patients with multiple ureteral calculi
* Patients whose urinary tracts are anatomically deformed or stenosed
* Patients who underwent invasive operations on their ureters before
* Patients whose blood creatinine levels are 2mg/dL and over
* Patients who are hypersensitive to silodosin
* Patients who take part in clinical trials other than this one
* Patients judged to be inappropriate for this clinical trial by investigators

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Actual)
Dates: Start 2011-10; Primary Completion 2012-03 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Expulsion rate of stones | 4 weeks
  1 week, 2 weeks, 4 weeks to visit and inspected. (Last visit four weeks) Results when the exhaust is used.

SECONDARY OUTCOMES:
Stone expulsion time | every 1 week or 2 weeks
Migration distance of stone | every 1 week or 2 weeks
Frequency of administration of oral or injectable analgesics | every 1 week or 2 weeks
Number of cases where subjects visited ER due to uncontrolled pains | every 1 week or 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Gwan-Joong Joo, Ph.D, Principal Investigator — Kangbuk Samsung Hospital; Tae-Yoong Jeong, Ph.D, Principal Investigator — Myongji Hospital; Young-Sik Kim, Ph.D, Principal Investigator — National Health Insurance Service Ilsan Hospital; Tak-Geun Yoo, Ph.D, Principal Investigator — Eulji Central Hospital; Jae-Yong Jeong, Ph.D, Principal Investigator — Inje University
Locations (5):
- South Korea (5):
  - NHIC Ilsan Hospital, Goyang-si, Gyonggi-Do
  - Myongji Hospital, Goyang-si, Gyonggi-Do
  - Kangbuk Samsung Medical Center, Seoul, Seoul
  - Inje Univ. Sanggye Paik Hospital, Seoul, Seoul
  - Eulji General Hospital, Seoul, Seoul